CLINICAL TRIAL: NCT06030297
Title: Diode Laser as a Biomarker for Neuropathic Pain of Peripheral Origin.
Acronym: DLss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Utah (Other)
Collaborators: Stanford University (Other); National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Rob Singleton, Professor and Vice Chair of Neurology, University of Utah
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: DLss-R61/R33
Record Dates: First submitted 2023-08-04; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Peripheral Neuropathy
Keywords: Biomarker; neuropathic pain; response biomarker
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neuralgia | interventions — Lidocaine; Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Response biomarker set-up and optimization in Healthy Subjects Examination of the relationship between Response Biomarker measures and severity of neuropathic pain in patients with peripheral neuropathy.
  Evaluate the the Response Biomarker using lidocaine patch as a peripherally acting neuropathic pain agents
Who Masked: Participant, Investigator
Masking Description: Unblinded team member will dispense patch masked to patient and investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Biomarker Optimization (Stanford) (Experimental): Screening for neuropathy, foot problems and diabetes Diode laser testing of C:Aδ ratio Non-invasive speckle imaging Quantitative sensory testing ZTlido 1.8% lidocaine patch testing in some subjects
  Interventions: Procedure: Diode Laser fiber type Selective Stimulator; Diagnostic Test: PeriCam PSI NR; Diagnostic Test: Medoc Quantitative Sensory Testing
- Neuropathy assessment and biomarker testing (Utah) (Experimental): History, physical, and neurological exam Nerve conduction study Medical record review of neuropathy history PROMIS pain severity and interference testing Brief pain inventory Norfolk quality of life questionnaire Quantitative sensory testing 3mm skin punch biopsy Diode laser testing of C:Aδ ratio Non-invasive speckle imaging
  Interventions: Procedure: Diode Laser fiber type Selective Stimulator; Diagnostic Test: PeriCam PSI NR; Diagnostic Test: Medoc Quantitative Sensory Testing
- Crossover testing in participants with painful neuropathy (ZTlido 1.8% lidocaine patch) (Active Comparator): History, physical, and neurological exam Nerve conduction study Medical record review of neuropathy history PROMIS pain severity and interference testing Brief pain inventory Norfolk quality of life questionnaire Quantitative sensory testing 3mm skin punch biopsy Diode laser testing of C:Aδ ratio Non-invasive speckle imaging ZTlido 1.8% lidocaine patch application to both feet for 7 days up to 12 hours per day.
  Interventions: Procedure: Diode Laser fiber type Selective Stimulator; Drug: ZTlido 1.8 % Topical System; Diagnostic Test: PeriCam PSI NR; Diagnostic Test: Medoc Quantitative Sensory Testing
- Crossover testing in participants with painful neuropathy (placebo patch) (Placebo Comparator): History, physical, and neurological exam Nerve conduction study Medical record review of neuropathy history PROMIS pain severity and interference testing Brief pain inventory Norfolk quality of life questionnaire Quantitative sensory testing 3mm skin punch biopsy Diode laser testing of C:Aδ ratio Non-invasive speckle imaging Placebo patch application to both feet for 7 days up to 12 hours per day.
  Interventions: Procedure: Diode Laser fiber type Selective Stimulator; Diagnostic Test: PeriCam PSI NR; Diagnostic Test: Medoc Quantitative Sensory Testing; Other: Inactive Topical System

INTERVENTIONS:
Procedure: Diode Laser fiber type Selective Stimulator — -Each patient will have an A and C fiber stimulation. Stimulation will be performed on the dorsum of the foot using stimulation previously published parameters to elicit "burning pain," which is from activation of C-fibers and "pinprick" pain from A-fib
  Other Names: DLss
Drug: ZTlido 1.8 % Topical System — ZTLI(diethylamino)-N-(2,6-dimethylphenyl), has an octanol:water partition ratio of 43 at pH 7.4. Each ZTLIDO contains 36 mg of lidocaine (18 mg per gram adhesive) in a non-aqueous base and also contains the following inactive ingredients: butylated hydroxytoluene, dipropylene glycol, isostearic acid, mineral oil, polyisobutylene, silicone dioxide, styrene/isoprene/styrene block copolymer, and terpene resin. DO (lidocaine topical system) 1.8% is a single-layer, drug-in-adhesive topical delivery system comprised of an adhesive material containing 36 mg lidocaine, which is applied to a pliable nonwoven cloth backing and covered with a polyethylene terephthalate film release liner. The release liner is removed prior to application to the skin. The size of ZTLIDO is 10 cm × 14 cm × 0.08 cm. Lidocaine, an amide local anesthetic, is chemically designated as acetamide, 2-
  Arms: Crossover testing in participants with painful neuropathy (ZTlido 1.8% lidocaine patch)
Diagnostic Test: PeriCam PSI NR — It is a method that visualizes tissue blood perfusion in real time. LASCA provides new means to study the microcirculation in ways that were not possible in the past. PeriCam PSI System combines dynamic response and high spatial resolution in one instrument, providing both real-time graphs and video recordings of the tissue being studied. To further enhance its usability, dedicated application software, PIMSoft, has been developed.
  Other Names: speckle imager
Diagnostic Test: Medoc Quantitative Sensory Testing — Quantitative sensory testing (QST) is a method through which sensory nerve function is quantitatively measured, based on responses of the subject. The peripheral sensory nervous system responds to specific stimuli of specific modality and intensity in a specific manner, which is well-known through many decades of research into human sensation. Thermal QST provides information about the function of small diameter unmyelinated (C fibers) and thinly myelinated (A-delta fibers) nerve fibers for which no nerve conduction test, or other objective tests exist.
  Small fiber nerve damage can manifest itself in thermal hypoesthesia (raised perception thresholds) or hyperalgesia (lowered pain thresholds).
  Other Names: QST
Other: Inactive Topical System — Inactive, non-medicated topical system comprised of an adhesive material containing, which is applied to a pliable nonwoven cloth backing and covered with a polyethylene terephthalate film release liner. The release liner is removed prior to application to the skin. The size of the system is 10 cm × 14 cm × 0.08 cm.
  Other Names: placebo patch
  Arms: Crossover testing in participants with painful neuropathy (placebo patch)

SUMMARY:
The R61 will perform a four-part double-blind randomized crossover study transitioning from a pretreatment baseline phase, to randomized treatment with either lidocaine or an identical placebo patch, washout, and alternate arm. DLss measures will be obtained before and after each phase. Twice daily report of pain using a visual analogue scale will track severity of ongoing spontaneous pain in participants. The hybrid biomarker will distinguish between placebo and active treatment arms, will significantly correlate with extent of neuropathic pain reduction during lidocaine, but will not change during the placebo phase or no-treatment lead-in. If preset Go/No-Go criteria are met, the subsequent R33 validation will then compare lidocaine patch and placebo treatment in a blinded, randomized parallel arm study.

DETAILED DESCRIPTION:
Pain caused by peripheral neuropathy is very common. Understanding patient response to pain and its treatment is one of the biggest barriers to development of effective medicines to reduce neuropathic pain. This project will develop and validate a non-invasive test that correlates with patients' experience of pain caused by peripheral neuropathy, a "pain biomarker". The biomarker device applies specialized light energy to skin on the top of the foot to selectively stimulate the nerve fibers in skin that sense and transmit pain. The test will determine how much energy is necessary to cause a person to feel the stimulus, or to first feel the pain of the stimulus. Sensory threshold to the stimulus, and transient enhancement of blood flow in the skin (flare) will be correlated with patient report of ongoing foot pain. Use of the experimental device, diagnostic testing, and use of lidocaine have risks that are explained in this document, but can include allergic reactions, discomfort, and temporary numbness.

SUMMARY OF STUDY PROCEDURES This study is being conducted by Drs. J. Robinson Singleton in the Department of Neurology at the University of Utah, and by Mikhail Nemenov PhD, of Stanford University, who developed the use of this technique for stimulating nerves in the skin. Study 1 will correlate the biomarker with patients' reported ongoing neuropathic foot. You may also be asked to participate in the Study 2, in which change in the biomarker will be correlated longitudinally to change in pain experience in a brief, randomized crossover trial of placebo or lidocaine patches applied to the top of the foot.

Optimization of DLss Biomarker in Healthy Subjects (Stanford)

Healthy subjects will be screened to exclude neuropathy, foot pain and diabetes then will have the DLss measures performed over several days. The visit lasts about 3-4 hours.

Study 1: biomarker correlation with ongoing pain (Utah)

This study consists of a single visit designed to evaluate possible neuropathy and assess its severity with history, standardized brief exam, and specialized testing. All participants will then rate their ongoing foot pain, and biomarker testing will be performed. The entire visit will take 2-3 hours. The purpose is to correlate the biomarker with patients reported ongoing neuropathic foot pain.

People with peripheral neuropathy. A total of 50 people will participate.

Study 2: biomarker correlation with change in pain during lidocaine treatment (Utah)

Study 2 is designed to see if change in neuropathic pain from treatment with an effective pain reducing agent correlates with change in the biomarker. Lidocaine, a locally acting anesthetic, will be applied to the top of the foot using a patch. The study is structured as a 4 week blinded and randomized crossover treatment trial and will five consist of 5 brief weekly study visits, once weekly over the 4 week study period. Crossover means that you will receive both treatments for a week each. Randomized means that the treatment you receive first, placebo or Lidocaine patch, will be chosen at random. Blinded means that you will not be told whether the treatment you receive during the treatment weeks is placebo or Lidocaine. The patches will look similar or identical. Neither you, nor the study coordinator will be able to tell the identity of the patches.

Study Segments: Each weekly segment of the study is proceeded and followed by a visit, in sequence. Each visit will include review of neuropathic pain and performance of QST and Biomarker Device assessment. There are four segments:

1. Baseline neuropathic pain evaluation. Each participant will be screened in clinic, then record daily pain severity for 7 days.
2. Treatment period 1. After this baseline period, each participant will be randomized to 7 days of treatment with a patch (either lidocaine or placebo) chosen by the study at random.
3. A 7-day wash out period without treatment.
4. Treatment period 2. Daily treatment with patch not received in the first treatment period.

A total of 44 people with neuropathy and associated neuropathic pain will participate

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Objective 1 (Stanford)

1. 18 -70 years of age
2. no complaints of peripheral neuropathy or other foot pain
3. no medical history of disease or medication use associated with peripheral neuropathy (e.g. diabetes)
4. no known allergy to lidocaine

Inclusion Criteria for Objective 2

1. . 18 years of age and older
2. Length dependent, sensory predominant, peripheral neuropathy from any non-acute acquired cause (e.g. diabetes, pre-diabetes, chemotherapy induced), OR musculoskeletal pain from plantar fasciitis or ankle sprain.

Inclusion Criteria for Objective 3

1. 18 years of age and older
2. Length dependent, sensory predominant, peripheral neuropathy from any non-acute acquired cause (e.g. diabetes, pre-diabetes, chemotherapy induced) .
3. Pain rating on Visual Analog Scale (VAS) > 30mm

Exclusion Criteria:

Exclusion criteria Objective 1 (Stanford)

1. complaints of peripheral neuropathy or other foot pain
2. medical history of disease or medication use associated with peripheral neuropathy (e.g. diabetes)
3. known allergy to lidocaine or other para-aminobenzioc acid derivative (ie: procaine, tetracaine, benzocaine)

Exclusion Criteria Objective 2 and 3

1. Acute peripheral neuropathy (e.g. Guillain Barre Syndrome, glucose correction neuropathy) because of concerns for stability of neuropathic pain over the period of study participation.
2. Bleeding diathesis, or history of severe bleeding with skin wounds.
3. known allergy to lidocaine or other para-aminobenzioc acid derivative (ie: procaine, tetracaine, benzocaine)

4. Taking exclusionary medications related to lidocaine, or with anti-arrhythmic properties, such as tocainide or mexilitine.

5. Severe liver disease

6. People currently receiving chemotherapy.

7. Unable to complete protocol requirements in the judgement of the investigator.-

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
CMi:Aδ ratio of amperage for sensory perception threshold following diode laser stimulation | 4 years
  Participants' will report sensory threshold and pain threshold following diode laser stimulation to foot dorsum of ascending power as measured by amperage.
Area of neurogenic flare response (mm squared) following repetitive subthreshold diode laser stimulation. | 24 months
  Foot dorsum skin will be repeatedly stimulated by diode laser and area of neurogenic flare measured using red blood cell reflectance using a speckle imager.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] FDA-NIH Biomarker Working Group. BEST (Biomarkers, EndpointS, and other Tools) Resource [Internet]. Silver Spring (MD): Food and Drug Administration (US); 2016-. Available from http://www.ncbi.nlm.nih.gov/books/NBK326791/ PMID 27010052
- [Background] DiBonaventura MD, Sadosky A, Concialdi K, Hopps M, Kudel I, Parsons B, Cappelleri JC, Hlavacek P, Alexander AH, Stacey BR, Markman JD, Farrar JT. The prevalence of probable neuropathic pain in the US: results from a multimodal general-population health survey. J Pain Res. 2017 Nov 1;10:2525-2538. doi: 10.2147/JPR.S127014. eCollection 2017. PMID 29138590
- [Background] Brix Finnerup N, Hein Sindrup S, Staehelin Jensen T. Management of painful neuropathies. Handb Clin Neurol. 2013;115:279-90. doi: 10.1016/B978-0-444-52902-2.00017-5. PMID 23931787
- [Background] Tracey I, Woolf CJ, Andrews NA. Composite Pain Biomarker Signatures for Objective Assessment and Effective Treatment. Neuron. 2019 Mar 6;101(5):783-800. doi: 10.1016/j.neuron.2019.02.019. PMID 30844399
- [Background] Davis KD, Aghaeepour N, Ahn AH, Angst MS, Borsook D, Brenton A, Burczynski ME, Crean C, Edwards R, Gaudilliere B, Hergenroeder GW, Iadarola MJ, Iyengar S, Jiang Y, Kong JT, Mackey S, Saab CY, Sang CN, Scholz J, Segerdahl M, Tracey I, Veasley C, Wang J, Wager TD, Wasan AD, Pelleymounter MA. Discovery and validation of biomarkers to aid the development of safe and effective pain therapeutics: challenges and opportunities. Nat Rev Neurol. 2020 Jul;16(7):381-400. doi: 10.1038/s41582-020-0362-2. Epub 2020 Jun 15. PMID 32541893
- [Background] Cuellar JM, Manering NA, Klukinov M, Nemenov MI, Yeomans DC. Thermal nociceptive properties of trigeminal afferent neurons in rats. Mol Pain. 2010 Jul 7;6:39. doi: 10.1186/1744-8069-6-39. PMID 20609212
- [Background] Veldhuijzen DS, Nemenov MI, Keaser M, Zhuo J, Gullapalli RP, Greenspan JD. Differential brain activation associated with laser-evoked burning and pricking pain: An event-related fMRI study. Pain. 2009 Jan;141(1-2):104-13. doi: 10.1016/j.pain.2008.10.027. Epub 2008 Dec 5. PMID 19058914
- [Background] Moeller-Bertram T, Schilling JM, Backonja MM, Nemenov MI. Sensory small fiber function differentially assessed with diode laser (DL) quantitative sensory testing (QST) in painful neuropathy (PN). Pain Med. 2013 Mar;14(3):417-21. doi: 10.1111/pme.12049. Epub 2013 Feb 22. PMID 23433028
- [Background] Rowbotham MC, Davies PS, Verkempinck C, Galer BS. Lidocaine patch: double-blind controlled study of a new treatment method for post-herpetic neuralgia. Pain. 1996 Apr;65(1):39-44. doi: 10.1016/0304-3959(95)00146-8. PMID 8826488
- [Background] Devers A, Galer BS. Topical lidocaine patch relieves a variety of neuropathic pain conditions: an open-label study. Clin J Pain. 2000 Sep;16(3):205-8. doi: 10.1097/00002508-200009000-00005. PMID 11014393
- [Background] Argoff CE. New analgesics for neuropathic pain: the lidocaine patch. Clin J Pain. 2000 Jun;16(2 Suppl):S62-6. doi: 10.1097/00002508-200006001-00011. PMID 10870742
- [Background] Katz NP, Gammaitoni AR, Davis MW, Dworkin RH; Lidoderm Patch Study Group. Lidocaine patch 5% reduces pain intensity and interference with quality of life in patients with postherpetic neuralgia: an effectiveness trial. Pain Med. 2002 Dec;3(4):324-32. doi: 10.1046/j.1526-4637.2002.02050.x. PMID 15099237
- [Background] Galer BS, Jensen MP, Ma T, Davies PS, Rowbotham MC. The lidocaine patch 5% effectively treats all neuropathic pain qualities: results of a randomized, double-blind, vehicle-controlled, 3-week efficacy study with use of the neuropathic pain scale. Clin J Pain. 2002 Sep-Oct;18(5):297-301. doi: 10.1097/00002508-200209000-00004. PMID 12218500
- [Background] Meier T, Wasner G, Faust M, Kuntzer T, Ochsner F, Hueppe M, Bogousslavsky J, Baron R. Efficacy of lidocaine patch 5% in the treatment of focal peripheral neuropathic pain syndromes: a randomized, double-blind, placebo-controlled study. Pain. 2003 Nov;106(1-2):151-8. doi: 10.1016/s0304-3959(03)00317-8. PMID 14581122
- [Background] Gammaitoni AR, Alvarez NA, Galer BS. Safety and tolerability of the lidocaine patch 5%, a targeted peripheral analgesic: a review of the literature. J Clin Pharmacol. 2003 Feb;43(2):111-7. doi: 10.1177/0091270002239817. PMID 12616661
- [Background] Kleggetveit IP, Namer B, Schmidt R, Helas T, Ruckel M, Orstavik K, Schmelz M, Jorum E. High spontaneous activity of C-nociceptors in painful polyneuropathy. Pain. 2012 Oct;153(10):2040-2047. doi: 10.1016/j.pain.2012.05.017. PMID 22986070
- [Background] Haroutounian S, Nikolajsen L, Bendtsen TF, Finnerup NB, Kristensen AD, Hasselstrom JB, Jensen TS. Primary afferent input critical for maintaining spontaneous pain in peripheral neuropathy. Pain. 2014 Jul;155(7):1272-1279. doi: 10.1016/j.pain.2014.03.022. Epub 2014 Apr 2. PMID 24704366
- [Background] Havlik RJ, Blackwelder WC, Kaslow R, Castelli W. Unlikely association between clinically apparent herpesvirus infection and coronary incidence at older ages. The Framingham Heart Study. Arteriosclerosis. 1989 Nov-Dec;9(6):877-80. doi: 10.1161/01.atv.9.6.877. PMID 2556099
- [Background] Schley M, Bayram A, Rukwied R, Dusch M, Konrad C, Benrath J, Geber C, Birklein F, Hagglof B, Sjogren N, Gee L, Albrecht PJ, Rice FL, Schmelz M. Skin innervation at different depths correlates with small fibre function but not with pain in neuropathic pain patients. Eur J Pain. 2012 Nov;16(10):1414-25. doi: 10.1002/j.1532-2149.2012.00157.x. Epub 2012 May 3. PMID 22556099
- [Background] Karlsson P, Hincker AM, Jensen TS, Freeman R, Haroutounian S. Structural, functional, and symptom relations in painful distal symmetric polyneuropathies: a systematic review. Pain. 2019 Feb;160(2):286-297. doi: 10.1097/j.pain.0000000000001381. PMID 30157133
- [Background] Schmelz M, Michael K, Weidner C, Schmidt R, Torebjork HE, Handwerker HO. Which nerve fibers mediate the axon reflex flare in human skin? Neuroreport. 2000 Feb 28;11(3):645-8. doi: 10.1097/00001756-200002280-00041. PMID 10718329
- [Background] Forstenpointner J, Naleschinski D, Wasner G, Hullemann P, Binder A, Baron R. Sensitized vasoactive C-nociceptors: key fibers in peripheral neuropathic pain. Pain Rep. 2019 Jan 18;4(1):e709. doi: 10.1097/PR9.0000000000000709. eCollection 2019 Jan-Feb. PMID 30801047
- [Background] Dworkin RH, Jensen MP, Gammaitoni AR, Olaleye DO, Galer BS. Symptom profiles differ in patients with neuropathic versus non-neuropathic pain. J Pain. 2007 Feb;8(2):118-26. doi: 10.1016/j.jpain.2006.06.005. Epub 2006 Sep 1. PMID 16949878
- [Background] Finnerup NB, Attal N, Haroutounian S, McNicol E, Baron R, Dworkin RH, Gilron I, Haanpaa M, Hansson P, Jensen TS, Kamerman PR, Lund K, Moore A, Raja SN, Rice AS, Rowbotham M, Sena E, Siddall P, Smith BH, Wallace M. Pharmacotherapy for neuropathic pain in adults: a systematic review and meta-analysis. Lancet Neurol. 2015 Feb;14(2):162-73. doi: 10.1016/S1474-4422(14)70251-0. Epub 2015 Jan 7. PMID 25575710
- [Background] Gudin J, Nalamachu S. Utility of lidocaine as a topical analgesic and improvements in patch delivery systems. Postgrad Med. 2020 Jan;132(1):28-36. doi: 10.1080/00325481.2019.1702296. Epub 2020 Jan 3. PMID 31900074
- [Background] Eriksson KF, Nilsson H, Lindgarde F, Osterlin S, Dahlin LB, Lilja B, Rosen I, Sundkvist G. Diabetes mellitus but not impaired glucose tolerance is associated with dysfunction in peripheral nerves. Diabet Med. 1994 Apr;11(3):279-85. doi: 10.1111/j.1464-5491.1994.tb00272.x. PMID 8033527
- [Background] Obrosova IG. Diabetic painful and insensate neuropathy: pathogenesis and potential treatments. Neurotherapeutics. 2009 Oct;6(4):638-47. doi: 10.1016/j.nurt.2009.07.004. PMID 19789069
- [Background] Stino AM, Smith AG. Peripheral neuropathy in prediabetes and the metabolic syndrome. J Diabetes Investig. 2017 Sep;8(5):646-655. doi: 10.1111/jdi.12650. Epub 2017 May 3. PMID 28267267
- [Background] Boger MS, Hulgan T, Haas DW, Mitchell V, Smith AG, Singleton JR, Peltier AC. Measures of small-fiber neuropathy in HIV infection. Auton Neurosci. 2012 Jul 2;169(1):56-61. doi: 10.1016/j.autneu.2012.04.001. Epub 2012 Apr 28. PMID 22542355
- [Background] Wulff EA, Wang AK, Simpson DM. HIV-associated peripheral neuropathy: epidemiology, pathophysiology and treatment. Drugs. 2000 Jun;59(6):1251-60. doi: 10.2165/00003495-200059060-00005. PMID 10882161
- [Background] Wolf S, Barton D, Kottschade L, Grothey A, Loprinzi C. Chemotherapy-induced peripheral neuropathy: prevention and treatment strategies. Eur J Cancer. 2008 Jul;44(11):1507-15. doi: 10.1016/j.ejca.2008.04.018. Epub 2008 Jun 18. PMID 18571399
- [Background] Windebank AJ, Grisold W. Chemotherapy-induced neuropathy. J Peripher Nerv Syst. 2008 Mar;13(1):27-46. doi: 10.1111/j.1529-8027.2008.00156.x. PMID 18346229
- [Background] Greene DA, Sima AA, Stevens MJ, Feldman EL, Lattimer SA. Complications: neuropathy, pathogenetic considerations. Diabetes Care. 1992 Dec;15(12):1902-25. doi: 10.2337/diacare.15.12.1902. PMID 1464245
- [Background] Gorson KC, Ropper AH. Idiopathic distal small fiber neuropathy. Acta Neurol Scand. 1995 Nov;92(5):376-82. doi: 10.1111/j.1600-0404.1995.tb00150.x. PMID 8610490
- [Background] Novella SP, Inzucchi SE, Goldstein JM. The frequency of undiagnosed diabetes and impaired glucose tolerance in patients with idiopathic sensory neuropathy. Muscle Nerve. 2001 Sep;24(9):1229-31. doi: 10.1002/mus.1137. PMID 11494278
- [Background] Visser NA, Vrancken AF, van der Schouw YT, van den Berg LH, Notermans NC. Chronic idiopathic axonal polyneuropathy is associated with the metabolic syndrome. Diabetes Care. 2013 Apr;36(4):817-22. doi: 10.2337/dc12-0469. Epub 2012 Nov 30. PMID 23204246
- [Background] Colloca L, Ludman T, Bouhassira D, Baron R, Dickenson AH, Yarnitsky D, Freeman R, Truini A, Attal N, Finnerup NB, Eccleston C, Kalso E, Bennett DL, Dworkin RH, Raja SN. Neuropathic pain. Nat Rev Dis Primers. 2017 Feb 16;3:17002. doi: 10.1038/nrdp.2017.2. PMID 28205574
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Bhupathiraju SN, Hu FB. Epidemiology of Obesity and Diabetes and Their Cardiovascular Complications. Circ Res. 2016 May 27;118(11):1723-35. doi: 10.1161/CIRCRESAHA.115.306825. PMID 27230638
- [Background] O'Connor AB. Neuropathic pain: quality-of-life impact, costs and cost effectiveness of therapy. Pharmacoeconomics. 2009;27(2):95-112. doi: 10.2165/00019053-200927020-00002. PMID 19254044
- [Background] Peltier A, Goutman SA, Callaghan BC. Painful diabetic neuropathy. BMJ. 2014 May 6;348:g1799. doi: 10.1136/bmj.g1799. PMID 24803311
- [Background] Tavee J, Zhou L. Small fiber neuropathy: A burning problem. Cleve Clin J Med. 2009 May;76(5):297-305. doi: 10.3949/ccjm.76a.08070. PMID 19414545
- [Background] McCarberg BH, Billington R. Consequences of neuropathic pain: quality-of-life issues and associated costs. Am J Manag Care. 2006 Jun;12(9 Suppl):S263-8. PMID 16774458
- [Background] Stewart WF, Ricci JA, Chee E, Hirsch AG, Brandenburg NA. Lost productive time and costs due to diabetes and diabetic neuropathic pain in the US workforce. J Occup Environ Med. 2007 Jun;49(6):672-9. doi: 10.1097/JOM.0b013e318065b83a. PMID 17563611
- [Background] Callaghan BC, Reynolds E, Banerjee M, Kerber KA, Skolarus LE, Burke JF. Longitudinal pattern of pain medication utilization in peripheral neuropathy patients. Pain. 2019 Mar;160(3):592-599. doi: 10.1097/j.pain.0000000000001439. PMID 30418352
- [Background] Mu A, Weinberg E, Moulin DE, Clarke H. Pharmacologic management of chronic neuropathic pain: Review of the Canadian Pain Society consensus statement. Can Fam Physician. 2017 Nov;63(11):844-852. PMID 29138154
- [Background] Lind AL, Wu D, Freyhult E, Bodolea C, Ekegren T, Larsson A, Gustafsson MG, Katila L, Bergquist J, Gordh T, Landegren U, Kamali-Moghaddam M. A Multiplex Protein Panel Applied to Cerebrospinal Fluid Reveals Three New Biomarker Candidates in ALS but None in Neuropathic Pain Patients. PLoS One. 2016 Feb 25;11(2):e0149821. doi: 10.1371/journal.pone.0149821. eCollection 2016. PMID 26914813
- [Background] Nwagwu CD, Sarris C, Tao YX, Mammis A. Biomarkers for Chronic Neuropathic Pain and their Potential Application in Spinal Cord Stimulation: A Review. Transl Perioper Pain Med. 2016;1(3):33-38. PMID 28480314
- [Background] Backryd E. Pain in the Blood? Envisioning Mechanism-Based Diagnoses and Biomarkers in Clinical Pain Medicine. Diagnostics (Basel). 2015 Mar 17;5(1):84-95. doi: 10.3390/diagnostics5010084. PMID 26854144
- [Background] Campbell JN, Meyer RA. Mechanisms of neuropathic pain. Neuron. 2006 Oct 5;52(1):77-92. doi: 10.1016/j.neuron.2006.09.021. PMID 17015228
- [Background] von Hehn CA, Baron R, Woolf CJ. Deconstructing the neuropathic pain phenotype to reveal neural mechanisms. Neuron. 2012 Feb 23;73(4):638-52. doi: 10.1016/j.neuron.2012.02.008. PMID 22365541
- [Background] van der Miesen MM, Lindquist MA, Wager TD. Neuroimaging-based biomarkers for pain: state of the field and current directions. Pain Rep. 2019 Aug 7;4(4):e751. doi: 10.1097/PR9.0000000000000751. eCollection 2019 Jul-Aug. PMID 31579847
- [Background] Leiser SC, Dunlop J, Bowlby MR, Devilbiss DM. Aligning strategies for using EEG as a surrogate biomarker: a review of preclinical and clinical research. Biochem Pharmacol. 2011 Jun 15;81(12):1408-21. doi: 10.1016/j.bcp.2010.10.002. Epub 2010 Oct 19. PMID 20937262
- [Background] Najib U, Bashir S, Edwards D, Rotenberg A, Pascual-Leone A. Transcranial brain stimulation: clinical applications and future directions. Neurosurg Clin N Am. 2011 Apr;22(2):233-51, ix. doi: 10.1016/j.nec.2011.01.002. PMID 21435574
- [Background] Pereira MP, Muhl S, Pogatzki-Zahn EM, Agelopoulos K, Stander S. Intraepidermal Nerve Fiber Density: Diagnostic and Therapeutic Relevance in the Management of Chronic Pruritus: a Review. Dermatol Ther (Heidelb). 2016 Dec;6(4):509-517. doi: 10.1007/s13555-016-0146-1. Epub 2016 Oct 11. PMID 27730494
- [Background] Smith AG, Lessard M, Reyna S, Doudova M, Singleton JR. The diagnostic utility of Sudoscan for distal symmetric peripheral neuropathy. J Diabetes Complications. 2014 Jul-Aug;28(4):511-6. doi: 10.1016/j.jdiacomp.2014.02.013. Epub 2014 Mar 6. PMID 24661818
- [Background] Singleton JR, Marcus RL, Lessard MK, Jackson JE, Smith AG. Supervised exercise improves cutaneous reinnervation capacity in metabolic syndrome patients. Ann Neurol. 2015 Jan;77(1):146-53. doi: 10.1002/ana.24310. Epub 2014 Dec 4. PMID 25388934
- [Background] Singleton JR, Marcus RL, Jackson JE, K Lessard M, Graham TE, Smith AG. Exercise increases cutaneous nerve density in diabetic patients without neuropathy. Ann Clin Transl Neurol. 2014 Oct;1(10):844-9. doi: 10.1002/acn3.125. Epub 2014 Oct 12. PMID 25493275
- [Background] Kalliomaki M, Kieseritzky JV, Schmidt R, Hagglof B, Karlsten R, Sjogren N, Albrecht P, Gee L, Rice F, Wiig M, Schmelz M, Gordh T. Structural and functional differences between neuropathy with and without pain? Exp Neurol. 2011 Oct;231(2):199-206. doi: 10.1016/j.expneurol.2011.05.019. Epub 2011 Jun 13. PMID 21683699
- [Background] Schmelz M, Schmidt R. Microneurographic single-unit recordings to assess receptive properties of afferent human C-fibers. Neurosci Lett. 2010 Feb 19;470(3):158-61. doi: 10.1016/j.neulet.2009.05.064. Epub 2009 May 28. PMID 19481585
- [Background] Donadio V, Liguori R. Microneurographic recording from unmyelinated nerve fibers in neurological disorders: an update. Clin Neurophysiol. 2015 Mar;126(3):437-45. doi: 10.1016/j.clinph.2014.10.009. Epub 2014 Oct 17. PMID 25457652
- [Background] Dubin AE, Patapoutian A. Nociceptors: the sensors of the pain pathway. J Clin Invest. 2010 Nov;120(11):3760-72. doi: 10.1172/JCI42843. Epub 2010 Nov 1. PMID 21041958
- [Background] Djouhri L, Koutsikou S, Fang X, McMullan S, Lawson SN. Spontaneous pain, both neuropathic and inflammatory, is related to frequency of spontaneous firing in intact C-fiber nociceptors. J Neurosci. 2006 Jan 25;26(4):1281-92. doi: 10.1523/JNEUROSCI.3388-05.2006. PMID 16436616
- [Background] Xiao WH, Bennett GJ. Chemotherapy-evoked neuropathic pain: Abnormal spontaneous discharge in A-fiber and C-fiber primary afferent neurons and its suppression by acetyl-L-carnitine. Pain. 2008 Apr;135(3):262-270. doi: 10.1016/j.pain.2007.06.001. Epub 2007 Jul 30. PMID 17659836
- [Background] Serra J, Bostock H, Sola R, Aleu J, Garcia E, Cokic B, Navarro X, Quiles C. Microneurographic identification of spontaneous activity in C-nociceptors in neuropathic pain states in humans and rats. Pain. 2012 Jan;153(1):42-55. doi: 10.1016/j.pain.2011.08.015. Epub 2011 Oct 10. PMID 21993185
- [Background] Bennett GJ, Liu GK, Xiao WH, Jin HW, Siau C. Terminal arbor degeneration--a novel lesion produced by the antineoplastic agent paclitaxel. Eur J Neurosci. 2011 May;33(9):1667-76. doi: 10.1111/j.1460-9568.2011.07652.x. Epub 2011 Mar 13. PMID 21395870
- [Background] Orstavik K, Namer B, Schmidt R, Schmelz M, Hilliges M, Weidner C, Carr RW, Handwerker H, Jorum E, Torebjork HE. Abnormal function of C-fibers in patients with diabetic neuropathy. J Neurosci. 2006 Nov 1;26(44):11287-94. doi: 10.1523/JNEUROSCI.2659-06.2006. PMID 17079656
- [Background] Schmidt R, Schmelz M, Weidner C, Handwerker HO, Torebjork HE. Innervation territories of mechano-insensitive C nociceptors in human skin. J Neurophysiol. 2002 Oct;88(4):1859-66. doi: 10.1152/jn.2002.88.4.1859. PMID 12364512
- [Background] Light AR. "Nocifensor" system re-revisited. Focus on "Two types of C nociceptor in human skin and their behavior in areas of capaicin-induced secondary hyperalgesia". J Neurophysiol. 2004 Jun;91(6):2401-3. doi: 10.1152/jn.00090.2004. No abstract available. PMID 15136601
- [Background] Lynn B, Schutterle S, Pierau FK. The vasodilator component of neurogenic inflammation is caused by a special subclass of heat-sensitive nociceptors in the skin of the pig. J Physiol. 1996 Jul 15;494 ( Pt 2)(Pt 2):587-93. doi: 10.1113/jphysiol.1996.sp021516. PMID 8842015
- [Background] Sauerstein K, Klede M, Hilliges M, Schmelz M. Electrically evoked neuropeptide release and neurogenic inflammation differ between rat and human skin. J Physiol. 2000 Dec 15;529 Pt 3(Pt 3):803-10. doi: 10.1111/j.1469-7793.2000.00803.x. PMID 11118507
- [Background] Mitchell K, Bates BD, Keller JM, Lopez M, Scholl L, Navarro J, Madian N, Haspel G, Nemenov MI, Iadarola MJ. Ablation of rat TRPV1-expressing Adelta/C-fibers with resiniferatoxin: analysis of withdrawal behaviors, recovery of function and molecular correlates. Mol Pain. 2010 Dec 17;6:94. doi: 10.1186/1744-8069-6-94. PMID 21167052
- [Background] Nolano M, Simone DA, Wendelschafer-Crabb G, Johnson T, Hazen E, Kennedy WR. Topical capsaicin in humans: parallel loss of epidermal nerve fibers and pain sensation. Pain. 1999 May;81(1-2):135-45. doi: 10.1016/s0304-3959(99)00007-x. PMID 10353501
- [Background] Lennertz RC, Medler KA, Bain JL, Wright DE, Stucky CL. Impaired sensory nerve function and axon morphology in mice with diabetic neuropathy. J Neurophysiol. 2011 Aug;106(2):905-14. doi: 10.1152/jn.01123.2010. Epub 2011 Jun 8. PMID 21653724
- [Background] Dyck PJ, Herrmann DN, Staff NP, Dyck PJ. Assessing decreased sensation and increased sensory phenomena in diabetic polyneuropathies. Diabetes. 2013 Nov;62(11):3677-86. doi: 10.2337/db13-0352. PMID 24158999
- [Background] Granovsky Y, Matre D, Sokolik A, Lorenz J, Casey KL. Thermoreceptive innervation of human glabrous and hairy skin: a contact heat evoked potential analysis. Pain. 2005 Jun;115(3):238-247. doi: 10.1016/j.pain.2005.02.017. Epub 2005 Apr 18. PMID 15911150
- [Background] Beydoun A, Dyke DB, Morrow TJ, Casey KL. Topical capsaicin selectively attenuates heat pain and A delta fiber-mediated laser-evoked potentials. Pain. 1996 May-Jun;65(2-3):189-96. doi: 10.1016/0304-3959(95)00161-1. PMID 8826506
- [Background] Bromm B, Treede RD. Nerve fibre discharges, cerebral potentials and sensations induced by CO2 laser stimulation. Hum Neurobiol. 1984;3(1):33-40. PMID 6330009
- [Background] Weidner C, Schmelz M, Schmidt R, Hansson B, Handwerker HO, Torebjork HE. Functional attributes discriminating mechano-insensitive and mechano-responsive C nociceptors in human skin. J Neurosci. 1999 Nov 15;19(22):10184-90. doi: 10.1523/JNEUROSCI.19-22-10184.1999. PMID 10559426
- [Background] Dusch M, Schley M, Rukwied R, Schmelz M. Rapid flare development evoked by current frequency-dependent stimulation analyzed by full-field laser perfusion imaging. Neuroreport. 2007 Jul 16;18(11):1101-5. doi: 10.1097/WNR.0b013e3281e72cff. PMID 17589307
- [Background] Treede RD, Meyer RA, Raja SN, Campbell JN. Evidence for two different heat transduction mechanisms in nociceptive primary afferents innervating monkey skin. J Physiol. 1995 Mar 15;483 ( Pt 3)(Pt 3):747-58. doi: 10.1113/jphysiol.1995.sp020619. PMID 7776255
- [Background] Tillman DB, Treede RD, Meyer RA, Campbell JN. Response of C fibre nociceptors in the anaesthetized monkey to heat stimuli: correlation with pain threshold in humans. J Physiol. 1995 Jun 15;485 ( Pt 3)(Pt 3):767-74. doi: 10.1113/jphysiol.1995.sp020767. PMID 7562615
- [Background] Greffrath W, Nemenov MI, Schwarz S, Baumgartner U, Vogel H, Arendt-Nielsen L, Treede RD. Inward currents in primary nociceptive neurons of the rat and pain sensations in humans elicited by infrared diode laser pulses. Pain. 2002 Sep;99(1-2):145-55. doi: 10.1016/s0304-3959(02)00071-4. PMID 12237192
- [Background] Brown JD, Saeed M, Do L, Braz J, Basbaum AI, Iadarola MJ, Wilson DM, Dillon WP. CT-guided injection of a TRPV1 agonist around dorsal root ganglia decreases pain transmission in swine. Sci Transl Med. 2015 Sep 16;7(305):305ra145. doi: 10.1126/scitranslmed.aac6589. PMID 26378245
- [Background] Fillingim RB, Loeser JD, Baron R, Edwards RR. Assessment of Chronic Pain: Domains, Methods, and Mechanisms. J Pain. 2016 Sep;17(9 Suppl):T10-20. doi: 10.1016/j.jpain.2015.08.010. PMID 27586827
- [Background] Younger J, McCue R, Mackey S. Pain outcomes: a brief review of instruments and techniques. Curr Pain Headache Rep. 2009 Feb;13(1):39-43. doi: 10.1007/s11916-009-0009-x. PMID 19126370
- [Background] Pickering G, Martin E, Tiberghien F, Delorme C, Mick G. Localized neuropathic pain: an expert consensus on local treatments. Drug Des Devel Ther. 2017 Sep 13;11:2709-2718. doi: 10.2147/DDDT.S142630. eCollection 2017. PMID 29066862
- [Background] Tzabazis A, Klyukinov M, Manering N, Nemenov MI, Shafer SL, Yeomans DC. Differential activation of trigeminal C or Adelta nociceptors by infrared diode laser in rats: behavioral evidence. Brain Res. 2005 Mar 10;1037(1-2):148-56. doi: 10.1016/j.brainres.2005.01.019. PMID 15777763
- [Background] Rage M, Van Acker N, Facer P, Shenoy R, Knaapen MW, Timmers M, Streffer J, Anand P, Meert T, Plaghki L. The time course of CO2 laser-evoked responses and of skin nerve fibre markers after topical capsaicin in human volunteers. Clin Neurophysiol. 2010 Aug;121(8):1256-66. doi: 10.1016/j.clinph.2010.02.159. Epub 2010 Mar 26. PMID 20347388
- [Background] Anand P, Bley K. Topical capsaicin for pain management: therapeutic potential and mechanisms of action of the new high-concentration capsaicin 8% patch. Br J Anaesth. 2011 Oct;107(4):490-502. doi: 10.1093/bja/aer260. Epub 2011 Aug 17. PMID 21852280
- [Background] Kennedy WR, Vanhove GF, Lu SP, Tobias J, Bley KR, Walk D, Wendelschafer-Crabb G, Simone DA, Selim MM. A randomized, controlled, open-label study of the long-term effects of NGX-4010, a high-concentration capsaicin patch, on epidermal nerve fiber density and sensory function in healthy volunteers. J Pain. 2010 Jun;11(6):579-87. doi: 10.1016/j.jpain.2009.09.019. Epub 2010 Apr 18. PMID 20400377
- [Background] Hovaguimian A, Gibbons CH. Diagnosis and treatment of pain in small-fiber neuropathy. Curr Pain Headache Rep. 2011 Jun;15(3):193-200. doi: 10.1007/s11916-011-0181-7. PMID 21286866
- [Background] Bhattacharya A, Wickenden AD, Chaplan SR. Sodium channel blockers for the treatment of neuropathic pain. Neurotherapeutics. 2009 Oct;6(4):663-78. doi: 10.1016/j.nurt.2009.08.001. PMID 19789071
- [Background] Manchikanti L, Helm S 2nd, Fellows B, Janata JW, Pampati V, Grider JS, Boswell MV. Opioid epidemic in the United States. Pain Physician. 2012 Jul;15(3 Suppl):ES9-38. PMID 22786464
- [Background] Rose MA, Kam PC. Gabapentin: pharmacology and its use in pain management. Anaesthesia. 2002 May;57(5):451-62. doi: 10.1046/j.0003-2409.2001.02399.x. PMID 11966555
- [Background] Colloca L. The Placebo Effect in Pain Therapies. Annu Rev Pharmacol Toxicol. 2019 Jan 6;59:191-211. doi: 10.1146/annurev-pharmtox-010818-021542. Epub 2018 Sep 14. PMID 30216744
- [Background] Raman R. Statistical methods in handling placebo effect. Int Rev Neurobiol. 2020;153:103-120. doi: 10.1016/bs.irn.2020.04.004. Epub 2020 Jun 9. PMID 32563284
- [Background] Bickel A, Kramer HH, Hilz MJ, Birklein F, Neundorfer B, Schmelz M. Assessment of the neurogenic flare reaction in small-fiber neuropathies. Neurology. 2002 Sep 24;59(6):917-9. doi: 10.1212/wnl.59.6.917. PMID 12297579
- [Background] Backonja MM, Attal N, Baron R, Bouhassira D, Drangholt M, Dyck PJ, Edwards RR, Freeman R, Gracely R, Haanpaa MH, Hansson P, Hatem SM, Krumova EK, Jensen TS, Maier C, Mick G, Rice AS, Rolke R, Treede RD, Serra J, Toelle T, Tugnoli V, Walk D, Walalce MS, Ware M, Yarnitsky D, Ziegler D. Value of quantitative sensory testing in neurological and pain disorders: NeuPSIG consensus. Pain. 2013 Sep;154(9):1807-1819. doi: 10.1016/j.pain.2013.05.047. Epub 2013 Jun 3. PMID 23742795
- [Background] Kirillova I, Teliban A, Gorodetskaya N, Grossmann L, Bartsch F, Rausch VH, Struck M, Tode J, Baron R, Janig W. Effect of local and intravenous lidocaine on ongoing activity in injured afferent nerve fibers. Pain. 2011 Jul;152(7):1562-1571. doi: 10.1016/j.pain.2011.02.046. Epub 2011 Apr 6. PMID 21474243
- [Background] Obreja O, Hirth M, Turnquist B, Rukwied R, Ringkamp M, Schmelz M. The differential effects of two sodium channel modulators on the conductive properties of C-fibers in pig skin in vivo. Anesth Analg. 2012 Sep;115(3):560-71. doi: 10.1213/ANE.0b013e3182542843. Epub 2012 May 10. PMID 22575571
- [Background] Krumova EK, Zeller M, Westermann A, Maier C. Lidocaine patch (5%) produces a selective, but incomplete block of Adelta and C fibers. Pain. 2012 Feb;153(2):273-280. doi: 10.1016/j.pain.2011.08.020. Epub 2011 Oct 11. PMID 21995882
- [Background] Kankel J, Obreja O, Kleggetveit IP, Schmidt R, Jorum E, Schmelz M, Namer B. Differential effects of low dose lidocaine on C-fiber classes in humans. J Pain. 2012 Dec;13(12):1232-41. doi: 10.1016/j.jpain.2012.09.008. PMID 23182228
- [Background] Kodaira M, Inui K, Kakigi R. Evaluation of nociceptive Adelta- and C-fiber dysfunction with lidocaine using intraepidermal electrical stimulation. Clin Neurophysiol. 2014 Sep;125(9):1870-7. doi: 10.1016/j.clinph.2014.01.009. Epub 2014 Jan 28. PMID 24566074
- [Background] Zhang J, Cavanaugh DJ, Nemenov MI, Basbaum AI. The modality-specific contribution of peptidergic and non-peptidergic nociceptors is manifest at the level of dorsal horn nociresponsive neurons. J Physiol. 2013 Feb 15;591(4):1097-110. doi: 10.1113/jphysiol.2012.242115. Epub 2012 Dec 24. PMID 23266932
- [Background] Mitchell K, Lebovitz EE, Keller JM, Mannes AJ, Nemenov MI, Iadarola MJ. Nociception and inflammatory hyperalgesia evaluated in rodents using infrared laser stimulation after Trpv1 gene knockout or resiniferatoxin lesion. Pain. 2014 Apr;155(4):733-745. doi: 10.1016/j.pain.2014.01.007. Epub 2014 Jan 13. PMID 24434730
- [Background] Singleton JR, Bixby B, Russell JW, Feldman EL, Peltier A, Goldstein J, Howard J, Smith AG. The Utah Early Neuropathy Scale: a sensitive clinical scale for early sensory predominant neuropathy. J Peripher Nerv Syst. 2008 Sep;13(3):218-27. doi: 10.1111/j.1529-8027.2008.00180.x. PMID 18844788
- [Background] McCormack HM, Horne DJ, Sheather S. Clinical applications of visual analogue scales: a critical review. Psychol Med. 1988 Nov;18(4):1007-19. doi: 10.1017/s0033291700009934. PMID 3078045
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Safikhani S, Gries KS, Trudeau JJ, Reasner D, Rudell K, Coons SJ, Bush EN, Hanlon J, Abraham L, Vernon M. Response scale selection in adult pain measures: results from a literature review. J Patient Rep Outcomes. 2018 Sep 6;2:40. doi: 10.1186/s41687-018-0053-6. eCollection 2017. PMID 30238085
- [Background] Rose M, Bjorner JB, Gandek B, Bruce B, Fries JF, Ware JE Jr. The PROMIS Physical Function item bank was calibrated to a standardized metric and shown to improve measurement efficiency. J Clin Epidemiol. 2014 May;67(5):516-26. doi: 10.1016/j.jclinepi.2013.10.024. PMID 24698295
- [Background] Zelman DC, Gore M, Dukes E, Tai KS, Brandenburg N. Validation of a modified version of the brief pain inventory for painful diabetic peripheral neuropathy. J Pain Symptom Manage. 2005 Apr;29(4):401-10. doi: 10.1016/j.jpainsymman.2004.06.018. PMID 15857744
- [Background] Smith AG, Howard JR, Kroll R, Ramachandran P, Hauer P, Singleton JR, McArthur J. The reliability of skin biopsy with measurement of intraepidermal nerve fiber density. J Neurol Sci. 2005 Jan 15;228(1):65-9. doi: 10.1016/j.jns.2004.09.032. Epub 2004 Nov 5. PMID 15607212
- [Background] Fruhstorfer H, Lindblom U, Schmidt WC. Method for quantitative estimation of thermal thresholds in patients. J Neurol Neurosurg Psychiatry. 1976 Nov;39(11):1071-5. doi: 10.1136/jnnp.39.11.1071. PMID 188989
- [Background] Yarnitsky D, Sprecher E, Zaslansky R, Hemli JA. Heat pain thresholds: normative data and repeatability. Pain. 1995 Mar;60(3):329-32. doi: 10.1016/0304-3959(94)00132-x. PMID 7596629
- [Background] Persaud N, Strichartz GR. Micromolar lidocaine selectively blocks propagating ectopic impulses at a distance from their site of origin. Pain. 2002 Sep;99(1-2):333-40. doi: 10.1016/s0304-3959(02)00163-x. PMID 12237212
- [Background] Chevrier P, Vijayaragavan K, Chahine M. Differential modulation of Nav1.7 and Nav1.8 peripheral nerve sodium channels by the local anesthetic lidocaine. Br J Pharmacol. 2004 Jun;142(3):576-84. doi: 10.1038/sj.bjp.0705796. Epub 2004 May 17. PMID 15148257
- [Background] Hans GH, Robert DN, Van Maldeghem KN. Treatment of an acute severe central neuropathic pain syndrome by topical application of lidocaine 5% patch: a case report. Spinal Cord. 2008 Apr;46(4):311-3. doi: 10.1038/sj.sc.3102098. Epub 2007 Jul 3. PMID 17607309
- [Background] Patel BK, Wendlandt BN, Wolfe KS, Patel SB, Doman ER, Pohlman AS, Hall JB, Kress JP. Comparison of Two Lidocaine Administration Techniques on Perceived Pain From Bedside Procedures: A Randomized Clinical Trial. Chest. 2018 Oct;154(4):773-780. doi: 10.1016/j.chest.2018.04.018. Epub 2018 Apr 24. PMID 29698720
- [Background] Park CH, Jung SH, Han CG. Effect of intravenous lidocaine on the neuropathic pain of failed back surgery syndrome. Korean J Pain. 2012 Apr;25(2):94-8. doi: 10.3344/kjp.2012.25.2.94. Epub 2012 Apr 4. PMID 22514776
- [Background] Calderon E, Calderon-Seoane ME, Garcia-Hernandez R, Torres LM. 5% Lidocaine-medicated plaster for the treatment of chronic peripheral neuropathic pain: complex regional pain syndrome and other neuropathic conditions. J Pain Res. 2016 Oct 6;9:763-770. doi: 10.2147/JPR.S113517. eCollection 2016. PMID 27785090
- [Background] Mills EJ, Chan AW, Wu P, Vail A, Guyatt GH, Altman DG. Design, analysis, and presentation of crossover trials. Trials. 2009 Apr 30;10:27. doi: 10.1186/1745-6215-10-27. PMID 19405975
- [Background] Diehr P, Chen L, Patrick D, Feng Z, Yasui Y. Reliability, effect size, and responsiveness of health status measures in the design of randomized and cluster-randomized trials. Contemp Clin Trials. 2005 Feb;26(1):45-58. doi: 10.1016/j.cct.2004.11.014. Epub 2005 Jan 27. PMID 15837452
- [Background] Hofseth LJ. Getting rigorous with scientific rigor. Carcinogenesis. 2018 Jan 12;39(1):21-25. doi: 10.1093/carcin/bgx085. No abstract available. PMID 28968787
- [Background] Brooks KG, Kessler TL. Treatments for neuropathic pain. The Pharmaceutical Journal. 2017; 9(12). Epub 13 Sept 2017
- [Background] Fitridge R, Thompson M, editors. Mechanisms of Vascular Disease: A Reference Book for Vascular Specialists [Internet]. Adelaide (AU): University of Adelaide Press; 2011. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK534260/ PMID 30484990
- [Background] A. Smith ML, J. Singleton. The diagnostic utility of nerve conduction studies and skin biopsy for diabetic neuropathy (DPN): a Bayesian analysis (S42.007). Neurology. Apr 2015;84.
- [Background] Hulicius E. aKV. Semiconductor lasers for medical applications. Lasers for Medical Applications Diagnostics, Therapy and Surgery. Woodhead Publishing Series in Electronic and Optical Materials: Elsevier BV; 2013. p. 222-50.
- [Background] JM. B. Pain as Human Experience: An Anthropological Perspective. JAMA. 1993; 270(8):998-9. doi:10.1001/jama.1993.03510080104042.
- [Background] Control CfD. Non Opioid treatments for chronic pain: principles of chronic pain treatment.2019. Epub 6/12/2019.
- [Background] Nemenov MIN, B.; Schmidt, R.; Kleggetveit, I.P.; Backonja M.; E., Jorum E.; Schmelz M, editors. Heating of deeper skin layers might detect spontaneously active heat-sensitized nociceptors. Neuroscience; 2015; Chicago.
- [Background] Foster-Palmer, S.C, Singleton, J.R., Revere, C., Marcus, R.L., Shakeri, M., Castillo, A., Shafi, S. 34-LB: Reliability of the UENS for Primary Care Neuropathy Screening. Diabetes. 2020;69. doi: 10.2337/db20-34-LB.
- [Background] Schwarz GE. Estimating the dimension of a model. Annals of Statistics. 1978;6(2):461-4.
- [Background] Verbeke, G. Linear Mixed Models for Longitudinal Data. In: Linear Mixed Models in Practice. Lecture Notes in Statistics, vol 126. Springer, New York, NY. 1997; doi: 10.1007/978-1-4612-2294-1_3